CLINICAL TRIAL: NCT05290363
Title: The Role of IL-23 in Chronic Inflammatory Disease: Exploring the Cellular and Molecular Targets of IL-23 Signaling in Peripheral and Axial Spondyloarthritis
Acronym: SpA23
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Janssen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-087; 2021-A02801-40 (Other: ANSM)
Record Dates: First submitted 2022-02-25; First posted 2022-03-22 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Spondyloarthritis
Keywords: interleukin-23; anti-IL-23 therapy; immune response; Spondyloarthritis
MeSH Terms: conditions — Spondylarthritis | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Two groups are included Group 1: 60 patients with axial SpA Group 2 : 30 patients with SpA or psoriatic arthritis and peripheral joint involvement, with a medical decision to treat peripheral joint inflammation by arthrocentesis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with axial spondyloarthritis participating in the study (Experimental): People with axial spondylarthritis (60 participants),
  Interventions: Other: Blood sampling
- Patients with peripheral spondyloarthritis participating in the study (Experimental): People with peripheral spondylarthritis or psoriatic arthritis (30 participants).
  Interventions: Other: Blood sampling; Other: synovial aspiration

INTERVENTIONS:
Other: Blood sampling — A 51 mL blood sample will be collected during the study
Other: synovial aspiration — If synovial aspiration is required in standard care for patients with peripheral spondylarthritis. Medical waste product will be collected for the study
  Arms: Patients with peripheral spondyloarthritis participating in the study

SUMMARY:
This is a research study involving humans, of the interventional type with minimal risks and constraints (RIPH2). It is a multicentric, non randomized prospective study aiming to better understand the mechanisms of the response to anti-IL-23 biologics in Spondyloarthritis patients attending the rheumatology department of Cochin, Saint-Antoine, Henri-Mondor hospitals (APHP) and Maison-Blanche Hospital (Reims).

DETAILED DESCRIPTION:
The aim of this project is to improve our understanding of the role of IL-23 in the pathophysiology of axial SpA and peripheral SpA.

This objective is detailed in three specific aims:

1. Define the effects of IL-23 on gene expression and cytokine production in innate and adaptive T lymphocytes from patients with SpA, and correlate them with the patient's genotype;
2. Phenotypically characterize immune cell populations in peripheral blood and in synovial fluid from peripheral SpA patients and identify at the single cell level the cells expressing the IL-23 receptor and/or producing IL-17.

The study population to be included are patients affected by SpA, attended to in the Rheumatology Departments of Cochin Hospital, Saint-Antoine Hospital Henri-Mondor hospitals in Paris (APHP) and Maison-Blanche Hospital in Reims. Participants will be divided into two groups: Group 1 comprises patients diagnosed with axial SpA, Group 2 SpA patients with peripheral SpA or psoriatic arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Age : Adults (>18 years)
* Satisfying ASAS diagnostic criteria for SpA
* Patient has active disease, defined by the presence of active synovitis, tendinitis, or dactylitis or significant inflammatory pain of the spine, judged by the examining clinician to be due to SpA.
* Informed consent signed
* Beneficiary of health insurance, except for the AME

Only for patients of Group 1 • Patient is naïve to biological therapies

Only for patients of Group 2

* Patient is affected by peripheral SpA (ASAS criteria) or psoriatic arthritis, with inflammation of peripheral joints
* Patient requires aspiration, as part of standard care

Non inclusion criteria:

* Patient is minor
* Patient is pregnant or breastfeeding
* Patient is immunocompromised
* Patient has received biological therapy with 2 or more biologics
* Patient is receiving corticosteroid treatment > 10 mg per day
* Patient is under legal protection, curators, guardianship
* Patient refuses consent
* Previous history of alcoholism, drug addiction, psychological problems, severe concomitant conditions that could invalidate the patient's consent or limit the patient's compliance to the treatment protocol.
* Beneficiary of the AME

Only for group 1

• Patient has received biological therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-10-06 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Profiling of open chromatin regions | 4 years
  Profiling of open chromatin regions (ATAC seq) in T lymphocytes, cultured in the presence or absence of IL-23in order to define the effects of IL-23 on gene expression and cytokine production in innate and adaptive T lymphocytes from patients with SpA, and correlate them with the patient's genotype
Profiling of transcriptome | 4 years
  Profiling of the transcriptome (RNA-seq) in T lymphocytes, cultured in the presence or absence of IL-23in order to define the effects of IL-23 on gene expression and cytokine production in innate and adaptive T lymphocytes from patients with SpA, and correlate them with the patient's genotype
Profiling of the genome | 4 years
  Profiling of the genome (genotyping) in T lymphocytes, cultured in the presence or absence of IL-23in order to define the effects of IL-23 on gene expression and cytokine production in innate and adaptive T lymphocytes from patients with SpA, and correlate them with the patient's genotype
Profiling of cytokine expression | 4 years
  Profiling of cytokine expression (Proximity Extension Assay technology) in T lymphocytes, cultured in the presence or absence of IL-23 in order to define the effects of IL-23 on gene expression and cytokine production in innate and adaptive T lymphocytes from patients with SpA, and correlate them with the patient's genotype
Single cell transcriptome analysis | 4 years
  Single cell transcriptome analysis of cells from patients with peripheral SpA will be performed to characterize immune cell populations in peripheral blood and in synovial fluid and identify at the single cell level the cells expressing the IL-23 receptor and/or producing IL-17;

SECONDARY OUTCOMES:
Measure lymphocyte levels to explore the effects of anti-IL23 treatment on the immune responses of axSpA patients | 4 years
  Define the effects in vitro of IL-23 blockade on immune responses in the peripheral blood of axSpA patients, using whole blood culture assays to profile stimulated protein secretion and gene expression, in the presence or absence of IL-23 inhibitors.
  As this therapy is not employed for the treatment of axSpA, we will characterize the in vitro effects of anti-IL-23 blockade on the immune responses of patients with axSpA, by analysing gene expression and protein secretion in whole blood cultures in the presence or absence of anti-IL-23 treatment.
  We will isolate MAIT, γδ TCR+, CD4+CCR6+ and CD8+CCR6+ (enriched in IL-23R+) T cell populations from peripheral blood of psoriasis patients and stimulate them through the T cell receptor (TCR), in the presence or absence of IL-23.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Hôpital Henri-Mondor, AP-HP - Service de Rhumatologie, Créteil
  - Hôpital Cochin, AP-HP - Department of Dermatology B, Paris
  - Hôpital Saint-Antoine, AP-HP - Service de Rhumatologie, Paris
  - Hôpital Maison Blanche - Service de Rhumatologie, Reims